CLINICAL TRIAL: NCT06898554
Title: Cross-Education Effect of Structured Balance Training Program on Spinal and Supraspinal Control in Athletes With Chronic Ankle Instability
Brief Title: Spinal and Supraspinal Control in Chronic Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayca Yagcioglu (Other)
Collaborators: Yeditepe University (Other); Yeditepe University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ayca Yagcioglu, MSc, Yeditepe University
Organization: Yeditepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YeditepeU23
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-11

CONDITIONS: Ankle Injuries; Ankle Sprains
Keywords: ankle, joint instability, cross-education, rehabilitation
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stable Group (Experimental): The intervention will be applied to only the stable ankle of the athletes with unilateral chronic ankle instability.
  Interventions: Other: The structured balance training protocol
- Unstable Group (Experimental): The intervention will be applied to only the unstable ankle of the athletes with unilateral chronic ankle instability.
  Interventions: Other: The structured balance training protocol
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Other: The structured balance training protocol — The structured balance training protocol consists of 7 exercises including balance and hop stabilization exercises for athletes with chronic ankle instability.
  Arms: Stable Group; Unstable Group

SUMMARY:
Ankle sprains are common sports injuries that often lead to chronic ankle instability (CAI). Patients with CAI experience deficits in neuromuscular control (NMC), including proprioception and strength. It is believed that damage to the ankle's ligament mechanoreceptors and the peroneal nerve after the initial ankle sprain can cause alterations in NMC, resulting in postural control and dynamic joint stability dysfunction. Inflammation related to recurrent ankle sprains may also contribute to neuromuscular impairments. Evidence suggests that bilateral postural control deficits occur after an ankle sprain, suggesting alterations in the central nervous system (CNS). Rehabilitation for CAI has been shown to lead to bilateral improvements in NMC, potentially due to neural alterations at both the spinal and supraspinal levels. Cross-education, which refers to the muscular crossed effect of unilateral training, has also been proposed as a mechanism for improving contralateral strength in neurologically healthy individuals. While the exact mechanisms underlying cross-education are not yet fully understood, evidence suggests that it involves neural adaptations at both spinal and supraspinal levels. This study aims to investigate the cross-education effect of a 6-week, unilateral balance training on corticomotor excitability, motor neuron pool excitability, and static and dynamic balance in athletes with chronic ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being an athlete between the ages of 18-25,
* Being a player in a field team sport such as basketball, volleyball, and handball,
* Having a history of at least 2 significant grade II LAS diagnosed by a physician,
* Related inflammatory symptoms, "giving away" sensation, obtaining a score ≤25 from the Cumberland Ankle Instability Tool (CAIT),
* A score <90% for the activities of daily living subscale and <80% for the sport subscale from the Foot and Ankle Ability Measure,
* Recurrent episodes of LAS of the injured ankle which occurred within at least 12 months.

Exclusion Criteria:

* Acute injury of lower extremity musculoskeletal structures in the last three months,
* Orthopedic surgery in any of the lower extremities,
* Bilateral ankle instability,
* Vestibular or balance disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Proprioceptive-Stabilometric Assessment | at the baseline and end of the intervention, 8 weeks
  The Prokin PK 252 will be used for proprioceptive-stabilometric assessment of the lower extremities, incorporating static and dynamic evaluations. The sensorimotor assessment will include the monopodal controlled-load proprioceptive control test and its variant with total load. Participants will perform movements with one foot on the platform, with angular displacements converted into electrical impulses for data acquisition. Static balance will be assessed on a stable platform for 30 seconds per ankle under eyes-open and eyes-closed conditions. Dynamic balance will be measured on an unstable platform under the same conditions. Proprioception will be evaluated on an unstable platform for 90 seconds, guiding the platform through horizontal, diagonal, and circular patterns as per the test program.
Transcranial Magnetic Stimulation | at the baseline and end of the intervention, 8 weeks
  Transcranial Magnetic Stimulation (TMS), a non-invasive neurophysiological technique, will be used to assess motor cortical function. Corticomotor excitability will be evaluated using dual-cone coil TMS to examine adaptations following cross-training after unilateral training. TMS will induce corticospinal volleys of direct (D) and indirect (I) waves.
  The resting motor threshold (rMT), a biomarker of upper motor neuron function, will be recorded. EMG recordings will assess corticomotor excitability, with Ag/AgCl electrodes placed on the tibialis anterior, peroneus longus, and gastrocnemius medialis muscles, following SENIAM guidelines.
  Participants will be seated in a TMS chair, and the hotspot in the left primary motor cortex will be identified. The MEP amplitude will be assessed at 120% rMT with 10 repetitions, and latency will be recorded. A 15-minute rest will be observed between muscle tests.
Hoffman Reflex | at the baseline and end of the intervention, 8 weeks
  The H-reflex will be measured to assess motor neuron pool excitability within the spinal loop, aiming to explain the mechanism underlying bilateral adaptations. As a valuable tool for evaluating neurological function in athletes, the H-reflex will provide insights into neurophysiological changes.
  EMG signals will be pre-amplified and bandpass filtered between 30-300 Hz and recorded from the peroneus longus, tibialis anterior, and gastrocnemius medialis muscles. The tibial nerve will be stimulated using single 1 ms square-wave pulses applied over the popliteal fossa.
  The test sequence will be randomized between stable and unstable ankles, ensuring balanced measurements. H-reflex excitability will be assessed for both ankles before and after the protocol to determine neuromuscular adaptations.

SECONDARY OUTCOMES:
Cumberland Ankle Instability Tool | at the baseline and end of the intervention, 8 weeks
  Cumberland Ankle Instability Tool (CAIT) containing a 9-item 30-point scale is a valid and reliable questionnaire for distinguishing and measuring the severity of functional instability (FI). Clinically, CAIT is an effective tool for evaluating the severity of FI, monitoring progress, and measuring treatment outcomes. In researches, the CAIT provides the identification, objective definition, and comparison of more homogenous subject groups. Participants scoring 25 or higher are less likely to have FI, while participants scoring 25 or lower are more likely to have FI.
Foot and Ankle Ability Measure (FAAM) | at the baseline and end of the intervention, 8 weeks
  Foot and Ankle Ability Measure (FAAM) is a self-reported tool improved to assess the physical function of individuals with foot and ankle-related musculoskeletal disorders. The valid and reliable Turkish version of FAAM (FAAM-T) was used (intraclass correlation coefficient [ICC] = 0.97 for FAAM-ADL and 0.94 for the FAAM-S subscales), which is a 29-item questionnaire, including 21-item Activities of Daily Living (ADL) and 8-item Sports subscales. Each answer is scored on a 5-point Likert scale ranging from 0 to 4. The maximum score is 84 points for the ADL subscale and 32 points for the Sports subscale. The total score is calculated as a percentage score ranging from 0% to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Berrin Aktekin, MD, Professor, Principal Investigator — Yeditepe University Hospital; Feyza Şule Hantal, PHd, Principal Investigator — Yeditepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Yeditepe University Koşuyolu Hospital, Istanbul
  - Yeditepe University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided